CLINICAL TRIAL: NCT05630443
Title: Effects of Prone Position After Major Abdominal Surgery
Acronym: EPOS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Cecilia Engström-Mattisson, MD PhD Associated Professor, Vastra Gotaland Region
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2021-06877-01
Record Dates: First submitted 2022-06-03; First posted 2022-11-29 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Surgery; Complications, Postoperative; Lung Infection
Keywords: complications postoperative; lungcomplications; abdominal surgery; prone position
MeSH Terms: conditions — Postoperative Complications | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS (No Intervention): Ordinary ERAS treatment postoperatively without any prone position or voicetraining
- +prone position (Active Comparator): Ordinary ERAS treatment adding the prone position and voicetraining in short intervals
  Interventions: Procedure: prone position

INTERVENTIONS:
Procedure: prone position — Ordinary ERAS treatment postoperatvely adding the prone position and voicetraining
  Arms: +prone position

SUMMARY:
Evaluation of postoperative prone position after major abdominal surgery. A randomized clinical trial of 100+100 patients and further add a voice/speech/singing protocol.

DETAILED DESCRIPTION:
Evaluation of postoperative prone position after major abdominal surgery. A randomized clinical trial of 100+100 patients and further add a voice/speech/singing protocol.

The patients will be randomized to the standard ERAS-protocol, enhanced recovery after surgery with or without adding periods of prone position after surgery.

They will be followed by protocol both as a momentum effect (experimental study) on POD 2-5 and also POD 7.

The aim is evaluation of prone position in order to improve the ventilation and hopefully diminish the risk of for example pneumonia and thromboembolism.

Inclusion criteria Patients referred to the Department of Surgery for major abdominal surgery of the esophagus, gastric- or pancreas surgery aim to cure.

Exclusion criteria Patients unable to understand Swedish in writing or speaking, preoperatively unable to perform a prone position.

The participation is voluntary and demands an inform consent from the patient operated upon.

The primary outcome is oxygen saturation and lung complications after surgery.

The secondary outcome is measurement of lung volumes, patient experience (7th graded Lickert scale), days of hospital care, 30 days complications etc.

Further investigations are perioperative properties as BMI, other forms of surgery, etc., and continues measurement of blood pressure, respiration frequency, heartrate, tubes and drainages, postoperative analgesic, blood samples with signs of bleeding, inflammation, infection.

ELIGIBILITY:
Patients eligable for abdominal surgery aim to cure with:

Inclusion Criteria:

- malignancy of the esophagus, gastric- or pancreas

Exclusion Criteria:

-.not able to understand Swedish in writing or speaking

- preoperatively unable to perform a prone position

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxygen saturation measurement postoperatively | an average of (POD) Postoperative day 2-7
  Measurement during sitting position
Number of participants with treatment-related adverse events of postoperative lung and abdominal complications incl a CT scan for objective measurement | through study completion, an average of 1 year
  Adverse events like pneumonia, lungembolism, lungempyema, interventions pankreatitis
Number of participants with treatment-related adverse events of postoperative lung and abdominal complications | through study completion, an average of 1 year
  Pneumonia, Lung embolism, Empyema of the lung, pankreatitis

SECONDARY OUTCOMES:
Number of participants with treatment-related diminished lung volumes | through study completion, an average of 1 year
  Spirometric measurements of diminished lung volumes
Number of days of Hospital care | through study completion, an average of 1 year
  Days of inhouse treatment
Number of participants needing intervention | through study completion, an average of 1 year
  Treament intervention like antibiotics or other medical or interventional treatment

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Engstrom Mattisson, MD PhD, Principal Investigator — Dept of Surgery, Sahlgrenska University Hospital, Gothenburg University, Sweden
Locations (1):
- Dept of Surgery, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
The template is only shared with the two invesitagtors in this application.